CLINICAL TRIAL: NCT01997073
Title: Effect of One-Lung Ventilation on Respiratory Gas Heat Content
Brief Title: One Lung Ventilation
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 489455
Record Dates: First submitted 2013-11-01; First posted 2013-11-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Evaluate the Changes in Respiratory Heat Content During One Lung Ventilation
Keywords: Respiratory enthalpy; One Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aims: 1) Measure exhalation enthalpy in patients receiving conventional positive pressure ventilation during stable hemodynamic conditions. 2) Measure exhalation enthalpy in patients following change from two-lung ventilation to one-lung ventilation while minute ventilation remains constant.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgical procedures requiring one lung ventilation.

Exclusion Criteria:

* Age <18 years. Pregnancy. Prisoners. Planned pneumoperitoneum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effect of One-Lung Ventilation on Respiratory Gas Heat Content | One year.
  Changes in respiratory heat content during one-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Neal W. Fleming, M.D., Ph.D., Principal Investigator — Professor, Director, Cardiovascular and Thoracic Anesthesiology
Locations (1):
- UC Davis Health System, Sacramento, California, United States